CLINICAL TRIAL: NCT02950272
Title: Chinese Adolescent Registry for Diabetes (CARD) Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: CARD-QiluH
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Chinese Adolescents With Diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years

SUMMARY:
The CARD study is a observational study which includes Chinese adolescents with diabetes aged 18-30. The study aims to explore the status of disease treatment, self-management, the relationship between disease treatment and disease outcome in Chinese adolescents with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed diabetes
* aged 14-30
* signed the informed consent

Exclusion Criteria:

* taking part in other drug research
* gestational diabetes
* diagnosed with tumor or cardiovascular disease

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chinese adolescents with diabetes aged 14-30.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
cardiovascular events | six year

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China